CLINICAL TRIAL: NCT02284737
Title: A Prospective, Multi-center, Randomized Control Trial to Investigate the Efficacy of Pulmonary Artery Denervation to Improved Functional Capacity and Hemodynamics in Patients With Pulmonary Artery Hypertension
Brief Title: A Study to Investigate the Efficacy of PADN to Improved Functional Capacity and Hemodynamics in Patients With PAH
Acronym: PADN-PAH
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of subjects.
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Shaoliang Chen, MD, Vice President, Nanjing First Hospital, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FirstNanjingMU
Record Dates: First submitted 2014-10-28; First posted 2014-11-06 (Estimated); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Pulmonary arterial hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- PADN + sildenafil (Experimental): Two to three ablations at 1-15 W for 120 seconds at each point were performed in the distal bifurcation area of the main PA.
  Interventions: Procedure: PADN; Drug: Sildenafil
- sham PADN + sildenafil (Sham Comparator): The radiofrequency ablation catheter placed, no ablations.
  Interventions: Procedure: sham PADN; Drug: Sildenafil

INTERVENTIONS:
Procedure: PADN — Contrast pulmonary artery angiography is performed to localize the pulmonary artery bifurcation level and to calculate the PA diameter. Once the anatomy is deemed acceptable, the radiofrequency ablation catheter is introduced into the distal bifurcation area of the main PA. The catheter is then maneuvered within the PA to allow energy delivery to ensure that the electrodes are tightly in contact with the endovascular surface. Two to three ablations at 1-15 W for 120 seconds at each point were performed in the distal bifurcation area of the main PA.
  Other Names: Pulmonary artery denervation
  Arms: PADN + sildenafil
Procedure: sham PADN — The radiofrequency ablation catheter placed, no ablations for patients in the sham PADN group.
  Other Names: sham pulmonary artery denervation
  Arms: sham PADN + sildenafil
Drug: Sildenafil — Participants initially received 5 mg tadalafil for the first 2 weeks in the two groups. The tadalafil dose may have been up titrated to 40 mg after 2 weeks, with maximum effects being obtained. The up titrated of tadalafil to 40 mg was not mandatory if the investigator decided for tolerability reasons the participants should remain on 5 mg.
  Other Names: Viagra

SUMMARY:
Pulmonary arterial hypertension (PAH) is characterized by premature death mainly because of progressive and severe right ventricular failure. Target drugs are reported to be associated with significant improvement of clinical outcome for PAH patients. However, previous studies using those target drugs focused on the change of 6-minute walk distance (6MWD) and or hemodynamic responses. As 6MWD has weak correlation with clinical outcome (time to clinical worsening, TTCW), benefits from target drugs for PAH patients are not clear. We previously reported the safety and efficacy of pulmonary artery denervation (PADN) for treatment of PAH patients who were unresponsive to target drugs. Hence, we design the randomized study to identify the effect of PADN on PAH.

DETAILED DESCRIPTION:
The current study is designed as a multicenter, randomized and prospective study aiming to compare the effect of PADN on PAH patients. Based on the previous studies, the rate of pulmonary arterial hypertension (PAH)-related event was around 30% after 6-month treatment using target drugs. And our previous data showed that this PAH-related event at 6-month after PADN procedure was 15%. As a result, a total of 270 PAH patients was required, with 135 patients/per group at a ratio of 1:1 randomization. All patients underwent an 18F-DOPA PET/CT scan of pulmonary arteries and the heart, performed at basement.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures;
* Men and women 18 years and older;
* Group I PAH, defined as a mPAP≥25mmHg, PCWP<15mmHg and PVR[The PVR =(mPAP-PCWP)/CO]>3.0 Woods unit.

Exclusion Criteria:

General exclusion criteria:

* Pregnancy and breast feeding mother;
* Estimated life expectancy <12 months;
* Scheduled major surgery in the next 6 months;
* Inability to follow the protocol and comply with follow-up requirements or any other reason that the investigator feels would place the patient at increased risk;
* Previous enrolment in this study or treatment with an investigational drug or device under another study protocol in the past 30 days.

Procedural exclusion criteria:

* WHO group II, III, IV, V PH
* Severe Renal dysfunction (Ccr<30 ml/min)
* Blood platelet count<100,000/L
* Expected life span<6-month
* Systematical inflammation
* Malignant cancer(s)
* Tricuspid valve stenosis, Supra-pulmonary valve stenosis
* Allergic to studied drugs or metal materials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-11-28 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Pulmonary artery hypertension (PAH)- related events | Baseline to month 6
  Including all-cause death, lung transplantation, atrial septostomy, worsening of PAH, initiation of treatment with intravenous or subcutaneous prostacyclin

SECONDARY OUTCOMES:
6-minute walk distance | Baseline to month 6
  The 6-minute walk distance (6MWD) test was conducted according to the American Thoracic Society guidelines (ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med 2002; 166(1):111-117.).
Pulmonary arterial pressure | Baseline to month 6
  Pulmonary arterial pressure was obtained with a 7-F flow-directed Swan-Ganz catheter at end-expiration.
Right atrial pressure | Baseline to month 6
  Right atrial pressure was obtained with a 7-F flow-directed Swan-Ganz catheter at end-expiration.
Pulmonary Vascular Resistance | Baseline to month 6
  PVR=[mean pulmonary arterial pressure-pulmonary artery occlusion pressure] / cardiac output
Cardiac output | Baseline to month 6
  The amount of blood the heart pumps through the circulatory system in a minute. Measured by right heart catheterization.
Trans-pulmonary pressure gradient | Baseline to month 6
  The transpulmonary pressure gradient (TPG), defined by the difference between mean pulmonary arterial pressure (P(pa)) and left atrial pressure (P(la).
Diastolic pressure gradient | Baseline to month 6
  The diastolic pressure gradient (DPG), defined by the difference between mean pulmonary arterial pressure and PA occlusion pressure.
Pulmonary arterial compliance | Baseline to month 6
  Pulmonary arterial compliance was obtained with a 7-F flow-directed Swan-Ganz catheter.
Borg Dyspnea Index | Baseline to month 6
  Borg Dyspnea Index is a measure of perceived shortness of breath: 0 units on a scale (none) to 10 units on a scale (maximum breathlessness).
World Health Organization (WHO) Functional Class | Baseline to month 6
  WHO Classes: I) pulmonary hypertension (PH); ordinary physical activity not limited or causes increased dyspnea, fatigue, chest pain, or presyncope. II) PH; ordinary physical activity mildly limited and causes increased dyspnea, fatigue, chest pain, or presyncope; comfortable at rest. III) PH; physical activity markedly limited and less than ordinary physical activity causes increased dyspnea, fatigue, chest pain, or presyncope; comfortable at rest. IV) PH; physical activity causes symptoms; signs of right heart failure; dyspnea/fatigue possible at rest.
New York functional class | Baseline to month 6
  NYHA Classes: I) Patients with no limitation of activities; they suffer no symptoms from ordinary activities. II) Patients with slight, mild limitation of activity; they are comfortable with rest or with mild exertion. III) Patients with marked limitation of activity; they are comfortable at rest. IV) Patients who should be at complete rest, confined to bed or chair; any physical activity brings on discomfort and symptoms occur at rest.

OTHER OUTCOMES:
Pulmonary artery perforation | During PADN procedure
  Number of Participants with pulmonary artery perforation
Pulmonary embolism | 6 months
  PE is classified by suspected and fatal ones. Suspected PE is defined as one of the following: 1) new intra-luminal filling defect on CT scan, MRI scan, or pulmonary angiogram; 2)new perfusion defect of at least 75% on V/Q lung scan; and 3) inconclusive spiral CT, pulmonary angiography or lung scan with demonstration of deep vein thrombosis in the lower extremities by venography. Fatal PE is PE based on objective diagnostic testing or autopsy or death not attributed to a documented cause and for which deep vein thrombosis/PE cannot be ruled out.
The prognostic role of 18F-DOPA PET/CT in patients with PAH | 6 months
  the prognostic role of 18F-DOPA PET/CT in patients with PAH.

CONTACTS AND LOCATIONS:
Overall Officials: Shao-Liang Chen, MD, Principal Investigator — Nanjing First Hospital, Nanjing Medical University, China
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen SL, Zhang FF, Xu J, Xie DJ, Zhou L, Nguyen T, Stone GW. Pulmonary artery denervation to treat pulmonary arterial hypertension: the single-center, prospective, first-in-man PADN-1 study (first-in-man pulmonary artery denervation for treatment of pulmonary artery hypertension). J Am Coll Cardiol. 2013 Sep 17;62(12):1092-1100. doi: 10.1016/j.jacc.2013.05.075. Epub 2013 Jul 10. PMID 23850902
- [Background] Chen SL, Zhang YJ, Zhou L, Xie DJ, Zhang FF, Jia HB, Wong SS, Kwan TW. Percutaneous pulmonary artery denervation completely abolishes experimental pulmonary arterial hypertension in vivo. EuroIntervention. 2013 Jun 22;9(2):269-76. doi: 10.4244/EIJV9I2A43. PMID 23466961